CLINICAL TRIAL: NCT07222982
Title: Social Groups for Autistic Young Adults (SDARI)
Brief Title: Social Groups for Autistic Young Adults (SDARIYA)
Acronym: SDARIYA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Matthew Lerner, Principal Investigator, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2409010784
Record Dates: First submitted 2025-10-01; First posted 2025-10-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; intervention; social performance
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: SDARIYA vs AYA (control)
Masking Description: N/A participants, providers and PI will know what condition the individual is placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDARI-YA (Experimental): follow SDARI Protocol
  Interventions: Behavioral: SDARI-YA
- AYA (Active Comparator): follow AYA Protocol
  Interventions: Other: AYA

INTERVENTIONS:
Behavioral: SDARI-YA — SDARI is a group-based, performance-based intervention designed to provide participants with opportunities to engage in and experience targeted interpersonal interactions, with minimal didactic instruction or instrumental reinforcement. The intervention consists of three core components:
  SDARI utilizes affectively motivating acting games that are adapted for the developmental stage and characteristics of the target population.
  Clinicians promote strong relationships among participants and between participants and clinicians by fostering a supportive and enjoyable environment, facilitating both structured and unstructured interactions, encouraging collaborative problem-solving, and reinforcing positive peer engagement.
  SDARI incorporates motivating activities-such as noncompetitive physical games, shared interests, and goal-oriented tasks-to enhance interpersonal motivation and engagement.
  Arms: SDARI-YA
Other: AYA — This group provides concrete presentation of thematic content and connects those themes to specific semi-structured, naturalistic games and activities. Themes are addressed and targeted according to the developmental needs of individual group members.
  Core Program Principles include:
  Use of recreational, motivational activities adapted for the target age range and population Positive reinforcement of interpersonal engagement through structured activities Integration of strong, age-appropriate motivators
  The AYA program uniquely combines these elements to facilitate both development and enjoyment. Group members engage in increasingly complex interpersonal interactions within the group setting and gain motivation to generalize these experiences across other environments, including home and educational contexts.
  Other Names: Control
  Arms: AYA

SUMMARY:
This is a clinical trial that will test whether a group program called SDARI (Socio-dramatic Affective Relational Intervention) can help autistic young adults between the ages of 18 and 30 feel more connected to others and improve their social relationships.

The study will try to answer:

Can SDARI be used successfully with autistic adults? Does SDARI help people feel more connected, supported, and mentally well?

There are two groups in the study. One group will participate in the SDARI program, and the other group will do different structured activities that don't focus on social connection. Researchers will compare the two groups to see if SDARI leads to better outcomes.

Participants will:

Complete screening to confirm eligibility (including autism traits and IQ) Attend weekly in-person group sessions for 10 weeks Take part in games and activities designed to support connection and collaboration Complete surveys and interviews before, during, and after the program Have the option to choose someone close to them (like a friend or family member) to fill out surveys about their experiences

DETAILED DESCRIPTION:
The proposed study will evaluate the Socio-dramatic Affective Relational Intervention (SDARI) in autistic young adults aged 18-30 years. SDARI is a group-based, performance-oriented intervention designed to support interpersonal engagement through structured, drama-based activities. The intervention emphasizes experiential learning and minimizes didactic instruction, focusing instead on affectively motivating games, collaborative interactions, and age-appropriate recreational activities.

Participants will be recruited through community organizations, university outreach channels, and autism service agencies. Eligibility will be determined through a multi-step screening process, including the RAADS, ADOS-2 Module 4, and KBIT-2R assessments. Eligible participants will be randomized into either the SDARI intervention group or a time-matched attention control group. Each group will meet weekly for 90-minute sessions over a 10-week period at the AJ Drexel Autism Institute.

The SDARI curriculum integrates three core components:

Use of improvisational and drama-based games tailored to the developmental stage and interests of autistic young adults.

Facilitation of peer-to-peer and participant-staff relationships to foster positive reinforcement and group cohesion.

Incorporation of motivating activities such as noncompetitive physical games and shared-interest tasks to enhance engagement.

The attention control condition will follow the same schedule and structure but will involve recreational activities that do not explicitly promote interpersonal interaction.

Participants will complete assessments at three timepoints: baseline (pre-intervention), post-intervention, and three-month follow-up. Measures will include self-report and informant-report questionnaires assessing interpersonal experiences, social networks, group cohesion, and mental health. Social Network Analysis (SNA) will be used to evaluate changes in participants' social connections and network structures over time.

All sessions will be video-recorded for fidelity monitoring. Staff will receive condition-specific training and weekly supervision to ensure consistency and adherence to the intervention protocol.

The study aims to assess the feasibility, acceptability, and preliminary efficacy of SDARI in autistic adult populations. Outcomes will inform future adaptations and dissemination of SDARI for broader use in clinical and community settings.

ELIGIBILITY:
Inclusion Criteria:

* Have graduated from high school (or an equivalent program) and are between the ages of 18-30 years old
* Demonstrate the ability to complete consent and all study measures and procedures in English
* Score ≥ 65 on the RAADS
* Score ≥ 70 on the KBIT-2R
* Score ≥ 6 on the ADOS-2 Module 4
* Are physically able to complete study activities (e.g., no significant physical impairment or mental condition restricting participation in study activities).
* Are physically able to travel to the AJ Drexel Autism Institute at Drexel University in Philadelphia, PA to attend all weekly study sessions

Exclusion Criteria:

* Are still enrolled in high school (or an equivalent program) or are not between the ages of 18-30 years old
* Are unable to complete study measures and/or procedures in English
* Are unable to complete consent procedures
* Score ≤ 65 on the RAADS
* Score ≤ 70 on the KBIT-2R
* Score ≤ 6 on the ADOS-2
* Cannot physically complete study activities
* Cannot physically travel to the AJ Drexel Autism Institute at Drexel University in Philadelphia, PA to attend study sessions
* Have a severe medical or psychiatric condition preventing them from safely completing study activities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Social Responsiveness | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by the Social Responsiveness Scale-2 (min= 0 and max=195), higher score= worse outcomes

SECONDARY OUTCOMES:
Friendship | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by the Quality of Socialization Questionnaire for Young Adults (QSQ-YA):
  For the conflict subscale (min 0, max= 24), a higher score indicates worse outcomes.
  For the frequency items (min 0, max n/a (i.e. questionnaire asks how many get togethers did you have in a week), a higher count of get-togethers or dates indicates better outcomes
Anxiety | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by Anxiety Scale for Autism (Adults) (ASA-A) (min=0, max=60, a higher score=worse outcomes)
Depression | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by The Patient Health Questionnaire (PHQ-9) (min=0, max=27, higher scores=worse outcomes)
Capacity for social and interpersonal pleasure | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) (min=17, max=102, higher scores indicate worse outcomes)
Cognitive flexibility | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by the Cognitive Flexibility Inventory (CFI) (min=20, max= 140, higher scores indicate better outcomes)
Loneliness | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  measured by the UCLA Loneliness Scale - Revised (min=20, max=80, higher score indicates worse outcomes.
Social processes/dimensions | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  Other informant report measured by the Stanford Social Dimensions Scale (SSDS) (Social Motivation (14 items): Scores range from 14 to 70.
  Social Affiliation (8 items): Scores range from 8 to 40. Expressive Social Communication (7 items): Scores range from 7 to 35. Social Recognition (7 items): Scores range from 7 to 35. Unusual Approach (4 items): Scores range from 4 to 20; higher scores indicate better outcomes)
Empathy | Day 1 (Baseline) Week 10 (Post-intervention) Week 22 (3-Month Follow-up)
  other informant report measured by the Toronto Empathy Questionnaire - Informant Version (TEQ-IV) (min=0, max=64, higher scores indicate better outcomes)
Group cohesion | Week 1, Week 3, Week 5, Week 7, Week 8, Week 10
  measured by the Group Cohesiveness Scale (GCS). (min=7 and max=35, higher scores indicate better outcomes)
Social networks | Day -14 to Day 0; Week 1 to Week 2; Week 11 to Week 12
  as measured by Social Networks Survey (SNS) (min/max scores= N/A)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lerner, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No